CLINICAL TRIAL: NCT02306733
Title: Ergometrine Versus Oxytocin in the Management of Atonic Post-partum Haemorrhage (PPH) in Women Delivered Vaginally: A Randomised Controlled Trial
Brief Title: Ergometrine Versus Oxytocin in the Management of Atonic Post-partum Haemorrhage (PPH) in Women Delivered Vaginally
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Lecturer of Gynecology and Obstetrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PPH 4
Record Dates: First submitted 2014-11-30; First posted 2014-12-03 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Post Partum Hemorrhage
Keywords: Post partum hemorrhage; Ergometrine; Oxytocin; Obstetrics
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Ergonovine; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ergometrine (Active Comparator): 100 women with atonic PPH will receive Ergometrine 400µgm (Methergin® Novartis, Switzerland) slowly intravenous (iv)
  Interventions: Drug: Ergometrine
- Oxytocin (Active Comparator): 100 women with atonic PPH will receive oxytocin 10 IU (Syntocinon® Novartis, Switzerland) slowly intravenous.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Ergometrine — 100 women with atonic PPH will receive Ergometrine 400µgm (Methergin® Novartis, Switzerland) slowly intravenous (iv).
  Arms: Ergometrine
Drug: Oxytocin — 100 women with atonic PPH will receive Oxytocin 10 IU(Syntocinon® Novartis, Switzerland) slowly intravenous. iv and group 2 will receive oxytocin
  Arms: Oxytocin

SUMMARY:
200 women with PPH will be randomly divided into 2 equal groups using computer generated random numbers. Group 1 will receive Ergometrine 400µgm (Methergin® Novartis, Switzerland) and group 2 will receive oxytocin 10 IU (Syntocinon®, Novartis, Switzerland). The investigators will not include a control group for ethical reasons.

DETAILED DESCRIPTION:
Obstetric haemorrhage remains one of the major causes of maternal death in both developed and developing countries. Postpartum haemorrhage (PPH) is defined as a blood loss >500 ml more of blood from the genital tract within 24 hours of the birth of a baby. PPH can be minor (500-1000 ml) or major (more than 1000 ml). The most frequent cause of PPH is uterine atony, contributing up to 80 % of the PPH cases.

Risk factors of atonic PPH include multiple pregnancy, placenta previa, previous PPH, body mass index (BMI) >30, prolonged labour, fetal macrosomia>4kg and primipara> 40 years.

Oxytocin is currently the uterotonic of first choice. It has proven to decrease the incidence of PPH by 40 % and has a rapid onset of action and a good safety profile. A disadvantage of oxytocin is its short half-life of 4-10 min, regularly requiring a continuous intravenous infusion or repeated intramuscular injections. Despite decades of empirical use in clinical practice, there are no trials comparing ergometrine and oxytocin as first-line agents for the treatment (rather than prevention) of PPH.

The study will be conducted in Cairo university hospitals and BeniSuef university hospitals. All patients attending the labour ward will be invited to participate in the study, the invitation will include a clear full explanation of the study. Only patients signing informed written consents will participate in the study.

200 women with PPH will be randomly divided into 2 equal groups using computer generated random numbers. Group 1 will receive Ergometrine 400µgm (Methergin® Novartis, Switzerland) and group 2 will receive oxytocin 10 IU (Syntocinon®, Novartis, Switzerland). The investigators will not include a control group for ethical reasons.

Once atonic PPH is diagnosed, 2 14-gauge cannulas will be inserted and a crystalloid intravenous (iv) infusion will be started. The allocated drug will be diluted in 10ml saline and will be given slowly iv, the fundus will be rubbed, A Foley's catheter will be inserted and a fluid balance chart will be commenced, pulse and blood pressure will be recorded every 15 minutes, venepuncture will be done for cross matching 4 units of blood, full blood count and coagulation screen.

The uterine tone and amount of bleeding will be noted and the need for further uterotonic agents will be determined 2 minutes after giving the drug. Blood loss will be estimated through weighing the swabs and using pictorial charts. Blood haemoglobin will be assessed 24 hours after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Atonic PPH

Exclusion Criteria:

* Gestational age<37 weeks
* Hypertension, cardiac disease or preeclampsia

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Need for other uterotonics | 2 minutes after giving the drug
  The uterus will be palpated to check the uterine tone and the amount of the bleeding will be estimated 2 minutes after giving the drug. Bleeding will be estimated by weighing the swaps and using pictorial charts.

SECONDARY OUTCOMES:
Development of major PPH | 10 minutes after giving the drug.
  Swaps will be weighed and pictorial charts will be used to estimate the amount of bleeding. Major PPH will be defined as bleeding >100ml.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - BeniSuef University hospitals, BeniSuef
  - Cairo university hospitals, Cairo

REFERENCES:
- [Background] Winter C, Macfarlane A, Deneux-Tharaux C, Zhang WH, Alexander S, Brocklehurst P, Bouvier-Colle MH, Prendiville W, Cararach V, van Roosmalen J, Berbik I, Klein M, Ayres-de-Campos D, Erkkola R, Chiechi LM, Langhoff-Roos J, Stray-Pedersen B, Troeger C. Variations in policies for management of the third stage of labour and the immediate management of postpartum haemorrhage in Europe. BJOG. 2007 Jul;114(7):845-54. doi: 10.1111/j.1471-0528.2007.01377.x. PMID 17567419
- [Background] Atukunda EC, Siedner MJ, Obua C, Mugyenyi GR, Twagirumukiza M, Agaba AG. Sublingual misoprostol versus intramuscular oxytocin for prevention of postpartum hemorrhage in Uganda: a double-blind randomized non-inferiority trial. PLoS Med. 2014 Nov 4;11(11):e1001752. doi: 10.1371/journal.pmed.1001752. eCollection 2014 Nov. PMID 25369200
- [Background] Ezeama CO, Eleje GU, Ezeama NN, Igwegbe AO, Ikechebelu JI, Ugboaja JO, Ezebialu IU, Eke AC. A comparison of prophylactic intramuscular ergometrine and oxytocin for women in the third stage of labor. Int J Gynaecol Obstet. 2014 Jan;124(1):67-71. doi: 10.1016/j.ijgo.2013.07.020. Epub 2013 Oct 5. PMID 24365208
- [Derived] Parry Smith WR, Papadopoulou A, Thomas E, Tobias A, Price MJ, Meher S, Alfirevic Z, Weeks AD, Hofmeyr GJ, Gulmezoglu AM, Widmer M, Oladapo OT, Vogel JP, Althabe F, Coomarasamy A, Gallos ID. Uterotonic agents for first-line treatment of postpartum haemorrhage: a network meta-analysis. Cochrane Database Syst Rev. 2020 Nov 24;11(11):CD012754. doi: 10.1002/14651858.CD012754.pub2. PMID 33232518